CLINICAL TRIAL: NCT06161831
Title: SEARCH II: Short Message Service (SMS) Electronic Adolescent Reminders for Completion of HPV Vaccination - Uganda: Randomized Controlled Trial
Brief Title: HPV Vaccine Reminders - SEARCH II Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Makerere University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Melissa Stockwell, Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: AAAT1572_2; R33CA253604 (NIH)
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Human Papillomavirus Vaccination
Keywords: Human papillomavirus; Vaccination; Text message; SMS; mHealth; Uganda

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Text message/automated phone reminders (Experimental): Text message or automated phone reminders
  Interventions: Behavioral: Text Message/automated phone reminder
- Usual Care (No Intervention): No reminders

INTERVENTIONS:
Behavioral: Text Message/automated phone reminder — Receipt of text message or automated phone reminders notifying when the next HPV vaccine dose is due (either first or second)
  Arms: Text message/automated phone reminders

SUMMARY:
This RCT will take place at health centres and their affiliated schools and community immunization centers overseen by the Kampala Capital City Authority (KCCA) as well as at the Makerere/Mulago/Columbia Adolescent Health Clinic in Kampala. The investigators will assess the impact of vaccine text message and automated phone reminders on human papillomavirus (HPV) vaccination initiation and completion.

DETAILED DESCRIPTION:
Cervical cancer is the leading female cancer in Uganda. HPV is the principal cause of cervical cancer. The national HPV vaccination program in Uganda includes preteen/ adolescent girls. Vaccinations are provided within schools or through community health centers. However, in Kampala, HPV vaccination especially series completion is low. While research regarding the use of text message vaccine reminders is strong in the U.S., their use has not been demonstrated in a preteen/adolescent population in Sub-Saharan Africa and other low and middle income countries (LMICs) in a full RCT. In this study, RCT caregivers of preteens/adolescents will be randomized and stratified by site, language and HPV vaccine dose needed (initiation vs. completion). Intervention families will receive text message or automated phone reminders based on family preference.

ELIGIBILITY:
Inclusion Criteria:

* Be a parenting adult of an adolescent girl aged 10-14 years
* Reside in Kampala and/or the surrounding districts
* Speak English or Luganda
* Have a cell phone with text messaging capability
* Must have ability to consent

Exclusion Criteria:

* Parenting adult speaks other language than English or Luganda only
* Parenting adult already enrolled in the study for another child
* Participation in previous HPV vaccine reminder study

Ages: 10 Years to 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 396 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to Receipt of First HPV Vaccine Dose | 12 months
  Timeliness of vaccination (time to event) will be measured
Time to Receipt of Second HPV Vaccine Dose | 12 months
  Timeliness of vaccination (time to event) will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Melissa S Stockwell, MD MPH, Principal Investigator — Columbia University
Locations (2):
- Columbia University Irving Medical Center, New York, New York, United States
- Makerere University/Mulago Hospital, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided